CLINICAL TRIAL: NCT06065124
Title: Bariatric Surgery Evaluation and Assessment of Treatment Efficacy in Heart Failure with Preserved Ejection Fraction - Intervention Trial
Brief Title: Bariatric Surgery Evaluation and Assessment of Treatment Efficacy - Intervention Trial
Acronym: BEAT-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEAT-IT trial
Record Dates: First submitted 2023-08-23; First posted 2023-10-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure with Preserved Ejection Fraction; Atrial Fibrillation
Keywords: Atrial Fibrillation; Heart Failure with Preserved Ejection Fraction; Bariatric surgery
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, randomized controlled, open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bariatric surgery strategy (Active Comparator): The intervention group will receive bariatric surgery including an intensive pre- and postoperative treatment scheme
  Interventions: Procedure: Bariatric surgery strategy
- Standard of Care (No Intervention): The control group will receive standard of care

INTERVENTIONS:
Procedure: Bariatric surgery strategy — Bariatric surgery including an intensive pre- and postoperative treatment scheme
  Arms: Bariatric surgery strategy

SUMMARY:
The goal of this clinical trial is to evaluate if a bariatric surgery strategy will improve clinical endpoints, cardiac parameters and functional status in patients with obesity (with BMI 32-40 kg/m2) and symptomatic HF with preserved or mildly reduced LVEF in combination with AF, as compared to standard of care. Patients will be randomized to either the Intervention group receiving bariatric surgery including an intensive pre- and postoperative treatment scheme or to the control group receiving standard of care.

DETAILED DESCRIPTION:
The primary objective is to study the effect of a bariatric surgery strategy on the hierarchical occurrence of: 1) all-cause mortality within 2 years, 2) emergency room visit or hospitalization for HF within 2 years, 3) recurrent ECG-documented AF within 2 years, 4) decrease of ≥30gr of left ventricular (LV) mass on transthoracic echocardiography, and 5) improvement of ≥5 points on the Kansas City Cardiomyopathy Questionnaire (KCCQ).

ELIGIBILITY:
Inclusion Criteria:

1. Signs and symptoms of HF according to the Europeans Society of Cardiology guideline;
2. Left ventricular ejection fraction ≥40%;
3. HFA-PEFF score ≥5 or HFA-PEFF score 2-4 in combination with positive stress test;
4. Between 45 and 70 years of age;
5. BMI 32-40 kg/m2;
6. Paroxysmal or persistent AF with a rhythm control strategy;
7. Willing to undergo both treatment strategies;
8. Written informed consent.

Exclusion Criteria:

1. BMI ≥40 kg/m2;
2. BMI <32 kg/m2;
3. Patients unwilling or unable to sign informed consent;
4. More than moderate mitral valve regurgitation/aortic valve regurgitation;
5. More than mild mitral valve stenosis/aortic valve stenosis;
6. Inadequate echocardiographic window for the assessment of LV mass index and/or the echocardiographic criteria needed for the HFA-PEFF score;
7. History of myocardial infarction, myocarditis, any invasive cardiac intervention (e.g. surgery, percutaneous coronary intervention, ablation) or stroke, <3 months before inclusion;
8. Scheduled for AF ablation;
9. Complex congenital heart disease;
10. Negative treatment advise from a specialized psychiatrist due to non-stabilized psychotic disorders, severe depression and/or personality disorders;
11. Patients unable to care for themselves or who are unable adapt to inherent lifestyle changes following bariatric surgery;
12. Any medical condition that limits life span <2 years;
13. Diseases requiring long term use of anti-inflammatory treatments;
14. The use of medication associated with substantial effects (>5 kg) on body weight.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Hierarchical endpoint | 2 years
  The hierarchical occurrence of: 1) All-cause mortality; 2) Emergency room visit or hospitalization for HF; 3) Recurrent ECG-documented AF; 4) Decrease of ≥30gr of LV mass on transthoracic echocardiography; 5) Improvement of ≥5 points on the Kansas City Cardiomyopathy Questionnaire (Scores are transformed to a range of 0-100, in which higher scores reflect better health status)

SECONDARY OUTCOMES:
All-cause mortality | 2 years
  All-cause mortality
Emergency room visit or hospitalization for HF | 2 years
  Emergency room visit or hospitalization for HF
Rate of recurrent AF | 2 years
  Recurrent AF documented on ECG
Decrease of left ventricular mass | 2 years
  Decrease of ≥30gr of LV mass measured by transthoracic echocardiography
Kansas City Cardiomyopathy Questionnaire improvement | 2 years
  Improvement of ≥5 points on the Kansas City Cardiomyopathy Questionnaire (scores are transformed to a range of 0-100, in which higher scores reflect better health status)

OTHER OUTCOMES:
Weight reduction | 2 years
  Measuring weight during clinical trial
Medication changes after surgery | 2 years
  Medication changes after surgery
Concomitant cardiovascular conditions and relevant comorbidities | 2 years
  Medical history of patient
Change in left atrial volume | 2 years
  Change in left atrial volume measured by transthoracic echocardiography
Change in left ventricular diastolic dysfunction | 2 years
  Change in left ventricular diastolic dysfunction measured by transthoracic echocardiography with the definition according to the leading guidelines
Change in left ventricular ejection fraction | 2 years
  Change in left ventricular ejection fraction measured by transthoracic echocardiography
Change in right ventricular function | 2 years
  Change in right ventricular function measured by transthoracic echocardiography with the definition according to the leading guidelines
Change in diameter of epicardial fat | 2 years
  Change in diameter of epicardial fat measured by transthoracic echocardiography
Healthcare resource use/costs | 2 years
  Measured with the iMedical Consumption Questionnaire (instrument for measuring medical consumption, costs will be estimated by given answers and relation to known costs of the items of medical consumption)
Health related quality of life / utility | 2 years
  Measured with the 5-level EQ-5D questionnaire (The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression)

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Rienstra, MD, PhD, Principal Investigator — University Medical Center Groningen; Dirk Jan van Veldhuisen, MD, PhD, Principal Investigator — University Medical Center Groningen; Thomas M Gorter, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - Rijnstate Hospital, Arnhem, Gelderland
  - University Medical Center Groningen, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: No